CLINICAL TRIAL: NCT02728323
Title: Ultrasound-guided Transversus Abdominis Plane Block in the Management of Acute Postoperative Pain Syndrome After Caesarean Section: a Double-blind Randomized Controlled Clinical Trial
Brief Title: Transversus Abdominis Plane Block in the Management of Acute Postoperative Pain Syndrome After Caesarean Section
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated
Sponsor: Emiliano Petrucci (Other)
Responsible Party: Sponsor-Investigator, Emiliano Petrucci, Anesthesist, San Salvatore Hospital of L'Aquila
Organization: San Salvatore Hospital of L'Aquila (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0057864/13
Record Dates: First submitted 2016-03-15; First posted 2016-04-05 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Levobupivacaine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levobupivacaine 100 mg, USG TAP Block (Active Comparator): 100 mg of Levobupivacaine by intramuscular injection, at the end of surgery
  Interventions: Drug: Levobupivacaine
- Placebo (Placebo Comparator): 20 ml of Saline (for 100 mg Levobupivacaine) intramuscularly, at the end of surgery
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Levobupivacaine — 100 mg of Levobupivacaine by intramuscular injection, at the end of surgery
  Other Names: Chirocaine
  Arms: Levobupivacaine 100 mg, USG TAP Block
Drug: Saline — 20 ml of saline saline by intramuscular injection, at the end of surgery
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
In many countries, caesarean section (CS) rates have been increasing. The international literature is unclear regarding the analgesic efficacy of the transversus abdominis plane block (TAPB) after a CS. In particular, no clinical trials exist in which the correct method of performing this block has been matched with the obtained analgesic effect after a CS. The primary goal of the study was to determine whether a correctly performed ultrasound-guided TAPB (USG-TAPB) could provide patients who underwent a CS with better control of acute postoperative pain during the first 72 hours after surgery

DETAILED DESCRIPTION:
Transversus abdominis plane block (TAPB) is a regional anesthetic technique that can provide analgesia for lower abdominal surgical procedures. Previous meta-analyses and recently published clinical trials have demonstrated promising results for this technique when it is used as part of multimodal postoperative pain treatment, but no consensus exists regarding the potency of this type of anesthetic procedure for analgesia after a CS. The primary goal of the study was to determine whether a correctly performed ultrasound-guided TAPB (USG-TAPB) could provide patients who underwent a CS with better control of acute postoperative pain during the first 72 hours after surgery. In this study, the correct execution of an USG-TAPB was verified, and then the procedure was matched with the obtained analgesic effect after a CS.

The secondary aims were to determine whether USG-TAPB could ensure a decline in postoperative requests for opiates and fewer opiate-related side effects, the return of faster bowel function, and shorter recovery time without generating critical hemodynamic changes.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* Caesarian Section. The Pfannenstiel incision was performed.

Exclusion Criteria:

* body mass index (BMI) >35
* allergy to local anesthetics
* skeletal and/or muscle abnormalities of the spine
* primary and/or secondary neurological diseases
* psychiatric diseases
* history of chronic pain and/or neuropathic disorders
* history of drug abuse
* state of sepsis
* infection and/or tumors within the skin on the back
* primary or secondary coagulopathies
* pre-eclampsia or eclampsia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain (Numeric Rate Scale) at 72 hours after surgery | 72 hours
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Patient satisfaction at 72 hours from surgery | 72 hours
  Descriptive scale of satisfaction in four step: not at all/slightly/somewhat/very satisfied)
The time of recovery of bowel function at 72 hours from surgery | 72 hours
  Time (in hours) to have defacation
The time of hospital discharge at 72 hours after surgery | 72 hours
  Time (days after surgery) for hospital discharging
The consumption of painkillers at 72 hours after surgery | 72 hours
  The equianalgesic dose (in mg) of morphine.
The healing of the surgical wound at 72 hours | 72 hours
  Descriptive scale of four step: unacceptable/acceptable/excellent healing

CONTACTS AND LOCATIONS:
Overall Officials: Pierfrancesco Fusco, MD, Principal Investigator — Anesthesia and Intensive care Unit, San Salvatore Academic Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fusco P, Cofini V, Petrucci E, Scimia P, Pozone T, Paladini G, Carta G, Necozione S, Borghi B, Marinangeli F. Transversus Abdominis Plane Block in the Management of Acute Postoperative Pain Syndrome after Caesarean Section: A Randomized Controlled Clinical Trial. Pain Physician. 2016 Nov-Dec;19(8):583-591. PMID 27906937